CLINICAL TRIAL: NCT01014650
Title: A Randomized, Double-Blind, Placebo-Controlled Single Intravenous Dose, Ascending Dose Level Study of the Safety, Tolerability and Pharmacokinetics of GLYX-13 in Normal Healthy Volunteers
Brief Title: Single Ascending Dose Safety, Tolerability and Pharmacokinetics Study of GLYX-13 in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GLYX13-C-101
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: glycine site partial agonist; normal volunteers; safety in normal volunteers
MeSH Terms: interventions — GLYX-13 peptide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV normal saline (Placebo Comparator): Single IV dose of normal saline as a control for safety and tolerability observations
  Interventions: Drug: IV normal saline
- IV GLYX-13 (Experimental): Single IV dose of GLYX-13
  Interventions: Drug: GLYX-13
- SC GLYX-13 (Experimental): Single SC dose
  Interventions: Drug: GLYX-13

INTERVENTIONS:
Drug: GLYX-13 — single IV or SC dose
  Other Names: NMDA receptor glycine site partial agonist
  Arms: IV GLYX-13; SC GLYX-13
Drug: IV normal saline — Single IV dose of normal saline
  Other Names: Saline
  Arms: IV normal saline

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of a single IV dose of GLYX-13, an N-Methyl-D-aspartate (NMDA) receptor glycine site functional partial agonist, in normal, healthy human volunteers.

DETAILED DESCRIPTION:
NMDA receptor glycine site partial agonists (GFPAs) have been demonstrated to be efficacious in animal models and/or in early human studies of several Central Nervous System (CNS) diseases including neuropathic pain, major depressive disorder, schizophrenia, Alzheimer's disease, anxiety including posttraumatic stress syndrome, and cognition in Down's syndrome and autism and others, without the psychomimetic side effects of NMDA receptor channel blockers. GLYX-13 has demonstrated a wide therapeutic ratio (500:1) between efficacy and side effects in animals. The purpose of this study is to evaluate the safety and pharmacokinetics of GLYX-13 following a single IV dose.

ELIGIBILITY:
Inclusion Criteria:

* clinical laboratory values < 2x the upper limit of normal
* ability to understand the requirements of the study and provide informed consent

Exclusion Criteria:

* alcohol abuse
* abuse of illicit substances
* current smoker
* currently taking prescription medications (other than for birth control)
* history of allergy to NMDA receptor ligands
* received another investigational drug within 30 days
* psychiatric disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Observed and laboratory-confirmed safety | four weeks

SECONDARY OUTCOMES:
Plasma concentration of parent drug will be assessed over time to estimate duration of pharmacodynamics in future efficacy trials. Plasma concentration and pharmacokinetics will be related in time to observed side effects. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Study Director — Lotus Clinical Research
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States

REFERENCES:
- [Derived] Preskorn S, Macaluso M, Mehra DO, Zammit G, Moskal JR, Burch RM; GLYX-13 Clinical Study Group. Randomized proof of concept trial of GLYX-13, an N-methyl-D-aspartate receptor glycine site partial agonist, in major depressive disorder nonresponsive to a previous antidepressant agent. J Psychiatr Pract. 2015 Mar;21(2):140-9. doi: 10.1097/01.pra.0000462606.17725.93. PMID 25782764